CLINICAL TRIAL: NCT05026333
Title: Pilot Study Aimed to Determine the Optimal Design for the UCLA/Danone Probiotic Intervention Study Related to Stress
Brief Title: Cognitive and Biological Responses in Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Arpana Gupta, Associate Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB # 20-001921
Record Dates: First submitted 2021-08-10; First posted 2021-08-30 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Stress, Psychological; Anxiety
Keywords: stress; women; high stress; low stress; perceived stress
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders | interventions — Phytoalexins

STUDY DESIGN:
Intervention Model Description: 2 groups (high stress/anxiety compared to low stress/anxiety) will be compared on their performance on within laboratory stress and cognitive tasks (4 different tests).
Who Masked: Participant
Masking Description: Participants will be blind to which stress/anxiety group they belong to. Researchers will not be blind to the group assignment as group assignment is part of the eligibility criteria for inclusion/enrollment in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Stress Group (Experimental): Group of high stress participants based on cutoff scores on the Perceived Stress Scale (PSS) and the STAI - State Anxiety Scale.
  Interventions: Other: Cognitive Stress Testing
- Low Stress Group (Experimental): Group of low stress participants based on cutoff scores on the Perceived Stress Scale (PSS) and the STAI - State Anxiety Scale.
  Interventions: Other: Cognitive Stress Testing

INTERVENTIONS:
Other: Cognitive Stress Testing — Cognitive and stress study with no product intervention and noninvasive. The high stress/anxiety group will be compared to the low stress/anxiety group in terms of changes from baseline to after the cognitive and stress tests (i.e., 4 laboratory tasks) and metabolite measures.
  Other Names: ANS testing; metabolites; cognitive tasks; stress tasks

SUMMARY:
The goal of this pilot part of the study (Step 1) is to identify the optimal population of high and low anxiety and stress individuals who will differentially respond to a laboratory stress task as measured by changes in subjective stress response (affect), cognition, attention, and biological measures (autonomic and metabolite responses).

Based on experience with different study populations, the investigator's believe that a healthy, homogenous population (Caucasian, women, premenopausal) with higher levels of state anxiety and perceived stress, and with greater responsiveness to laboratory stress tasks (which can also be used in the probiotic intervention study in Step 2) will provide the highest likelihood of identifying the underlying central mechanisms of stress responsiveness in Step 1 and then for the probiotic intervention in Step 2.

For this pilot study, the investigator's will look at baseline measures to determine differences in responses to four subjective (affect/cognition/attention) stress tasks (primary endpoints) and biological (secondary endpoints) measures in a high stress group and a low stress group.

If for Step 1 of the study, the investigator's are able to verify the stratification of the participants into high and low stress groups based on questionnaire data and show differences between participants with high and low perceived stress in psychological characteristics, lab stress tasks and potentially in biological responses, this will help to determine the optimal cut off values, and the optimal stress tasks to be conducted in the planned probiotic intervention study of Step 2.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Female
* 18-45 years of age
* For the high perceived stress group: a PSS score of 15 or higher and a STAI-S of 39 or higher
* For the low perceived stress group: a PSS score of 8 or lower and a STAI-S score of 24 or lower

Exclusion Criteria:

* Any ongoing major medical, psychological, or psychiatric conditions and recent changes (3mo) in the use of psychoactive medications or other medications that interfere with the measured outcomes.
* Medical conditions such as current neurological, cardiovascular, hepatic, renal, autoimmune diseases, diabetes, or cancer. This includes having a current or past within 1 year diagnosis of GI disorders, including but not limited to IBS, IBD, Celiac, or other nutritional deficiency/disease, current eating disorder, or past weight loss surgery.
* Psychological conditions such as anxiety and depression (I.e., without history of Diagnostic and Statistical Manual (DSM-4) psychiatric diagnosis.
* Prior/Concomitant Therapy (e.g., Recent changes in the use of psychoactive medications or other medications that interfere with the measured outcomes, as determined by the PI).
* Subject involved in any other clinical study within the preceding month or in the exclusion period after another clinical study.
* Positive test for COVID-19 infection in the past month or if presenting symptoms of COVID-19 infection in the past 2 weeks.

Diet:

* Participant who changes her dietary habits within the preceding 4 weeks.
* Participants on probiotics will be asked to wait 1 month before enrollment in the study.
* Participant with an eating disorder.
* Participant with special medicated diet (e.g., for obesity, anorexia, metabolic pathology).
* Participant under artificial nutrition in the last 1 month.
* Participant planning to modify her dietary habits during the course of the study.

Other Exclusions:

* Pregnant women or women planning to become pregnant during the study; breast-feeding women based on the interview at screen (Visit 1) and the urine test on day of stress test (Visit 2).
* Smoker with a moderate to high level of dependence to nicotine (e.g., more than 1/2 a pack of cigarettes a day).
* Participant consuming regularly more than 3 units of alcohol per day (1 unit = 10mL or 8g).
* Participants not able to answer questionnaires by writing, whatever the reason.
* Participant with loos of liberty, by administrative or judicial decision.
* Participant who is major but with a legal guardian.
* Participant on antibiotics will be asked to wait 3 months before enrollment in the study.

Medications not Authorized:

* Opiates/Narcotics
* Chronic/Daily use of analgesics
* Anti-seizure meds
* Antidepressants (5HT3's / Tricyclics etc.) are allowed as long as it's been a stable dose for 3 months
* Medications for ADD/ADHD (I.e., Adderall)
* Any medication for appetite suppression
* Chronic use of laxative/antidiarrheals/medications affecting GI motility
* Insulin
* Bile acid sequestrants
* Use of centrally acting medications that will interfere with CNS testing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Differences in Subjective Stress Response | Pre and Post laboratory testing during the in-clinic visit lasting 2-4 hours.
  Between group differences in pre-and post- of the "overall" negative and positive affect subscale scores from the Positive Affect and Negative Affect Scale (PANAS) administered at baseline immediately before and after the 4 brief and well validated laboratory stress tasks. PANAS scores can range from 10-50 for both the positive and negative affect, with the lower scores representing lower levels of positive/negative affect, and higher scores representing higher levels of positive/negative affect.

SECONDARY OUTCOMES:
Differences in Attention/Executive Function | Throughout the Color Stroop laboratory test at the in-clinic visit lasting approximately 30 minutes.
  Between and within group differences on the time it takes to complete the Color Stroop attention/executive function lab stress task.
Differences in Emotional Arousal System | Throughout the IAPS laboratory test during the in-clinic visit lasting approximately 30 minutes.
  Between and within group differences in valence and emotional arousal ratings during the IAPS task.
Differences in Subjective Stress Response | Pre and Post the arithmetic stress task during the in-clinic visit lasting approximately 30 minutes.
  Between and within group differences on the negative affect subscale from the Brief Positive Affect and Negative Affect Scale (PANAS) before and after the arithmetic task. PANAS scores can range from 10-50 for both the positive and negative affect, with the lower scores representing lower levels of positive/negative affect, and higher scores representing higher levels of positive/negative affect.
Changes in Autonomic Measures - Heart Rate Variability | Throughout each laboratory test during the in-clinic visit lasting 2-4 hours.
  Between and within group differences in overall average change in heart rate variability pre and post each laboratory stress task.
Differences in Attention/Executive Function | Throughout the Trails A & B laboratory tests at the in-clinic visit lasting approximately 30 minutes.
  Between and within group differences on the time it takes to complete the Trails A and B attention/executive function lab stress task.
Changes in Autonomic Measures - diastolic and systolic blood pressure | Throughout each laboratory test during the in-clinic visit lasting 2-4 hours.
  Between and within group differences in overall average change in both diastolic and systolic blood pressure pre and post each laboratory stress task.
Changes in Autonomic Measures - Skin Conductance | Throughout each laboratory test during the in-clinic visit lasting 2-4 hours.
  Between and within group differences in overall average change in skin conductance pre and post each laboratory stress task.

OTHER OUTCOMES:
Changes in Stress-Related Plasma Metabolite Concentrations as measured via a blood sample and processed by Ixcela for targeted stress-related metabolites. | Pre and Post laboratory testing during the in-clinic visit lasting 2-4 hours.
  Between and within group differences in pre- and post- laboratory stress tasks in targeted stress-related metabolite concentrations assessed with the Ixcela Panel and analyzed using a Welch's two-sample t-test to identify overall metabolite changes. Extensive literature details the role of metabolites in modulation of the brain, and widespread effects on excitatory neurotransmission and neuroinflammation. (Metabolites Targeted will include the following pathways: Tryptophan, Purine, Serotonin, Kynurenine, Hypoxanthine, Xanthosine, Xanthine, Guanosine, Guanine, Uric Acid, Methionine, 4-Hydroxy 3-Methoxy Phenylacetic Acid, DL 4-Hydroxy, 3-Methoxy Mandelic Acid, Methoxy Hydroxyphenyl, Glycol, 4HPLA, 2HPAC, 4HPAC).

CONTACTS AND LOCATIONS:
Overall Officials: Arpana Gupta, PhD, Principal Investigator — The Regents of the University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to make the de-identified data available for sharing with other researchers

REFERENCES:
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Berthoud HR. Interactions between the "cognitive" and "metabolic" brain in the control of food intake. Physiol Behav. 2007 Aug 15;91(5):486-98. doi: 10.1016/j.physbeh.2006.12.016. Epub 2007 Jan 12. PMID 17307205
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Murphy KJ, Hodges TE, Sheppard PAS, Troyer AK, Hampson E, Galea LAM. Sex differences in cortisol and memory following acute social stress in amnestic mild cognitive impairment. J Clin Exp Neuropsychol. 2020 Nov;42(9):881-901. doi: 10.1080/13803395.2020.1825633. Epub 2020 Oct 6. PMID 33023371
- [Background] Helminen EC, Morton ML, Wang Q, Felver JC. Stress Reactivity to the Trier Social Stress Test in Traditional and Virtual Environments: A Meta-Analytic Comparison. Psychosom Med. 2021 Apr 1;83(3):200-211. doi: 10.1097/PSY.0000000000000918. PMID 33534392
- [Background] Wheelock MD, Goodman AM, Harnett NG, Wood KH, Mrug S, Granger DA, Knight DC. Sex-related Differences in Stress Reactivity and Cingulum White Matter. Neuroscience. 2021 Apr 1;459:118-128. doi: 10.1016/j.neuroscience.2021.02.014. Epub 2021 Feb 13. PMID 33588003
- [Background] Olfert MD, Barr ML, Charlier CC, Greene GW, Zhou W, Colby SE. Sex Differences in Lifestyle Behaviors among U.S. College Freshmen. Int J Environ Res Public Health. 2019 Feb 7;16(3):482. doi: 10.3390/ijerph16030482. PMID 30736399
- [Background] Luque B, Castillo-Mayen R, Cuadrado E, Gutierrez-Domingo T, Rubio SJ, Arenas A, Delgado-Lista J, Perez Martinez P, Tabernero C. The Role of Emotional Regulation and Affective Balance on Health Perception in Cardiovascular Disease Patients According to Sex Differences. J Clin Med. 2020 Sep 30;9(10):3165. doi: 10.3390/jcm9103165. PMID 33007817
- [Background] Marin IA, Goertz JE, Ren T, Rich SS, Onengut-Gumuscu S, Farber E, Wu M, Overall CC, Kipnis J, Gaultier A. Microbiota alteration is associated with the development of stress-induced despair behavior. Sci Rep. 2017 Mar 7;7:43859. doi: 10.1038/srep43859. PMID 28266612
- [Background] Schneider TR, Rench TA, Lyons JB, Riffle RR. The influence of neuroticism, extraversion and openness on stress responses. Stress Health. 2012 Apr;28(2):102-10. doi: 10.1002/smi.1409. Epub 2011 Jun 15. PMID 22281953
- [Background] Cohen S, Janicki-Deverts D, Doyle WJ, Miller GE, Frank E, Rabin BS, Turner RB. Chronic stress, glucocorticoid receptor resistance, inflammation, and disease risk. Proc Natl Acad Sci U S A. 2012 Apr 17;109(16):5995-9. doi: 10.1073/pnas.1118355109. Epub 2012 Apr 2. PMID 22474371
- [Background] Villada C, Hidalgo V, Almela M, Salvador A. Individual Differences in the Psychobiological Response to Psychosocial Stress (Trier Social Stress Test): The Relevance of Trait Anxiety and Coping Styles. Stress Health. 2016 Apr;32(2):90-9. doi: 10.1002/smi.2582. Epub 2014 Jun 11. PMID 24916722
- [Background] Walter S, Kessler H, Gruss S, Jerg-Bretzke L, Scheck A, Strobel J, Hoffmann H, Traue HC. The influence of neuroticism and psychological symptoms on the assessment of images in three-dimensional emotion space. Psychosoc Med. 2011;8:Doc04. doi: 10.3205/psm000073. Epub 2011 Jun 6. PMID 21698089
- [Background] Crow AJD. Associations Between Neuroticism and Executive Function Outcomes: Response Inhibition and Sustained Attention on a Continuous Performance Test. Percept Mot Skills. 2019 Aug;126(4):623-638. doi: 10.1177/0031512519848221. Epub 2019 May 30. PMID 31146642
- [Background] Craske MG, Waters AM, Nazarian M, Mineka S, Zinbarg RE, Griffith JW, Naliboff B, Ornitz EM. Does neuroticism in adolescents moderate contextual and explicit threat cue modulation of the startle reflex? Biol Psychiatry. 2009 Feb 1;65(3):220-6. doi: 10.1016/j.biopsych.2008.07.020. Epub 2008 Sep 11. PMID 18789433
- [Background] Naliboff BD, Waters AM, Labus JS, Kilpatrick L, Craske MG, Chang L, Negoro H, Ibrahimovic H, Mayer EA, Ornitz E. Increased acoustic startle responses in IBS patients during abdominal and nonabdominal threat. Psychosom Med. 2008 Oct;70(8):920-7. doi: 10.1097/PSY.0b013e318186d858. Epub 2008 Oct 8. PMID 18842745
- [Background] Weng YJ, Gan HY, Li X, Huang Y, Li ZC, Deng HM, Chen SZ, Zhou Y, Wang LS, Han YP, Tan YF, Song YJ, Du ZM, Liu YY, Wang Y, Qin N, Bai Y, Yang RF, Bi YJ, Zhi FC. Correlation of diet, microbiota and metabolite networks in inflammatory bowel disease. J Dig Dis. 2019 Sep;20(9):447-459. doi: 10.1111/1751-2980.12795. Epub 2019 Aug 1. PMID 31240835
- [Background] Floegel A, Wientzek A, Bachlechner U, Jacobs S, Drogan D, Prehn C, Adamski J, Krumsiek J, Schulze MB, Pischon T, Boeing H. Linking diet, physical activity, cardiorespiratory fitness and obesity to serum metabolite networks: findings from a population-based study. Int J Obes (Lond). 2014 Nov;38(11):1388-96. doi: 10.1038/ijo.2014.39. Epub 2014 Mar 10. PMID 24608922
- [Background] Yamada T, Takahashi D, Hase K. The diet-microbiota-metabolite axis regulates the host physiology. J Biochem. 2016 Jul;160(1):1-10. doi: 10.1093/jb/mvw022. Epub 2016 Mar 11. PMID 26970281
- [Background] Rhee SH, Pothoulakis C, Mayer EA. Principles and clinical implications of the brain-gut-enteric microbiota axis. Nat Rev Gastroenterol Hepatol. 2009 May;6(5):306-14. doi: 10.1038/nrgastro.2009.35. PMID 19404271
- [Background] Galley JD, Bailey MT. Impact of stressor exposure on the interplay between commensal microbiota and host inflammation. Gut Microbes. 2014 May-Jun;5(3):390-6. doi: 10.4161/gmic.28683. Epub 2014 Apr 1. PMID 24690880
- [Background] Goyal N, Shukla G. Probiotic Lactobacillus rhamnosus GG modulates the mucosal immune response in Giardia intestinalis-infected BALB/c mice. Dig Dis Sci. 2013 May;58(5):1218-25. doi: 10.1007/s10620-012-2503-y. Epub 2012 Dec 21. PMID 23263901
- [Background] Thomas CM, Hong T, van Pijkeren JP, Hemarajata P, Trinh DV, Hu W, Britton RA, Kalkum M, Versalovic J. Histamine derived from probiotic Lactobacillus reuteri suppresses TNF via modulation of PKA and ERK signaling. PLoS One. 2012;7(2):e31951. doi: 10.1371/journal.pone.0031951. Epub 2012 Feb 22. PMID 22384111
- [Background] Schwarcz R, Bruno JP, Muchowski PJ, Wu HQ. Kynurenines in the mammalian brain: when physiology meets pathology. Nat Rev Neurosci. 2012 Jul;13(7):465-77. doi: 10.1038/nrn3257. PMID 22678511
- [Background] Bischoff SC, Barbara G, Buurman W, Ockhuizen T, Schulzke JD, Serino M, Tilg H, Watson A, Wells JM. Intestinal permeability--a new target for disease prevention and therapy. BMC Gastroenterol. 2014 Nov 18;14:189. doi: 10.1186/s12876-014-0189-7. PMID 25407511
- [Background] Clarke G, Fitzgerald P, Cryan JF, Cassidy EM, Quigley EM, Dinan TG. Tryptophan degradation in irritable bowel syndrome: evidence of indoleamine 2,3-dioxygenase activation in a male cohort. BMC Gastroenterol. 2009 Jan 20;9:6. doi: 10.1186/1471-230X-9-6. PMID 19154614
- [Background] Mawe GM, Hoffman JM. Serotonin signalling in the gut--functions, dysfunctions and therapeutic targets. Nat Rev Gastroenterol Hepatol. 2013 Aug;10(8):473-86. doi: 10.1038/nrgastro.2013.105. Epub 2013 Jun 25. PMID 23797870
- [Background] Gershon MD, Tack J. The serotonin signaling system: from basic understanding to drug development for functional GI disorders. Gastroenterology. 2007 Jan;132(1):397-414. doi: 10.1053/j.gastro.2006.11.002. PMID 17241888
- [Background] Elsenbruch S. How positive and negative expectations shape the experience of visceral pain. Handb Exp Pharmacol. 2014;225:97-119. doi: 10.1007/978-3-662-44519-8_6. PMID 25304528
- [Background] Aizawa E, Sato Y, Kochiyama T, Saito N, Izumiyama M, Morishita J, Kanazawa M, Shima K, Mushiake H, Hongo M, Fukudo S. Altered cognitive function of prefrontal cortex during error feedback in patients with irritable bowel syndrome, based on FMRI and dynamic causal modeling. Gastroenterology. 2012 Nov;143(5):1188-1198. doi: 10.1053/j.gastro.2012.07.104. Epub 2012 Jul 27. PMID 22841782
- [Background] Kennedy PJ, Clarke G, O'Neill A, Groeger JA, Quigley EM, Shanahan F, Cryan JF, Dinan TG. Cognitive performance in irritable bowel syndrome: evidence of a stress-related impairment in visuospatial memory. Psychol Med. 2014 May;44(7):1553-66. doi: 10.1017/S0033291713002171. Epub 2013 Aug 29. PMID 23985155
- [Background] Tanaka Y, Kanazawa M, Fukudo S, Drossman DA. Biopsychosocial model of irritable bowel syndrome. J Neurogastroenterol Motil. 2011 Apr;17(2):131-9. doi: 10.5056/jnm.2011.17.2.131. Epub 2011 Apr 27. PMID 21602989
- [Background] Renaud P, Blondin JP. The stress of Stroop performance: physiological and emotional responses to color-word interference, task pacing, and pacing speed. Int J Psychophysiol. 1997 Sep;27(2):87-97. doi: 10.1016/s0167-8760(97)00049-4. PMID 9342640
- [Background] Douchamps J. A brief, versatile, computerized, stress-inducing task derived from the Stroop color word test. Methods Find Exp Clin Pharmacol. 1988 Sep;10(9):595-601. PMID 3226226
- [Background] Sugg MJ, McDonald JE. Time course of inhibition in color-response and word-response versions of the Stroop task. J Exp Psychol Hum Percept Perform. 1994 Jun;20(3):647-75. doi: 10.1037//0096-1523.20.3.647. PMID 8027716
- [Background] Corrigan JD, Hinkeldey NS. Relationships between parts A and B of the Trail Making Test. J Clin Psychol. 1987 Jul;43(4):402-9. doi: 10.1002/1097-4679(198707)43:43.0.co;2-e. PMID 3611374
- [Background] Gaudino EA, Geisler MW, Squires NK. Construct validity in the Trail Making Test: what makes Part B harder? J Clin Exp Neuropsychol. 1995 Aug;17(4):529-35. doi: 10.1080/01688639508405143. PMID 7593473
- [Background] Mikels JA, Fredrickson BL, Larkin GR, Lindberg CM, Maglio SJ, Reuter-Lorenz PA. Emotional category data on images from the International Affective Picture System. Behav Res Methods. 2005 Nov;37(4):626-30. doi: 10.3758/bf03192732. PMID 16629294
- [Background] Wei M, Roodenrys S, Miller L, Barkus E. Complex Scenes From the International Affective Picture System (IAPS). Exp Psychol. 2020 May;67(3):194-201. doi: 10.1027/1618-3169/a000488. PMID 32900297
- [Background] Constantinescu AC, Wolters M, Moore A, MacPherson SE. A cluster-based approach to selecting representative stimuli from the International Affective Picture System (IAPS) database. Behav Res Methods. 2017 Jun;49(3):896-912. doi: 10.3758/s13428-016-0750-0. PMID 27287449
- [Background] Armario P, del Rey RH, Martin-Baranera M, Almendros MC, Ceresuela LM, Pardell H. Blood pressure reactivity to mental stress task as a determinant of sustained hypertension after 5 years of follow-up. J Hum Hypertens. 2003 Mar;17(3):181-6. doi: 10.1038/sj.jhh.1001530. PMID 12624608
- [Background] Henze GI, Zankert S, Urschler DF, Hiltl TJ, Kudielka BM, Pruessner JC, Wust S. Testing the ecological validity of the Trier Social Stress Test: Association with real-life exam stress. Psychoneuroendocrinology. 2017 Jan;75:52-55. doi: 10.1016/j.psyneuen.2016.10.002. Epub 2016 Oct 17. PMID 27771565
- [Background] Naliboff BD, Benton D, Solomon GF, Morley JE, Fahey JL, Bloom ET, Makinodan T, Gilmore SL. Immunological changes in young and old adults during brief laboratory stress. Psychosom Med. 1991 Mar-Apr;53(2):121-32. doi: 10.1097/00006842-199103000-00002. PMID 2031066
- [Background] Thayer JF, Ahs F, Fredrikson M, Sollers JJ 3rd, Wager TD. A meta-analysis of heart rate variability and neuroimaging studies: implications for heart rate variability as a marker of stress and health. Neurosci Biobehav Rev. 2012 Feb;36(2):747-56. doi: 10.1016/j.neubiorev.2011.11.009. Epub 2011 Dec 8. PMID 22178086
- [Background] Ahluwalia N, Dwyer J, Terry A, Moshfegh A, Johnson C. Update on NHANES Dietary Data: Focus on Collection, Release, Analytical Considerations, and Uses to Inform Public Policy. Adv Nutr. 2016 Jan 15;7(1):121-34. doi: 10.3945/an.115.009258. Print 2016 Jan. PMID 26773020
- [Background] Crawford JR, Henry JD. The positive and negative affect schedule (PANAS): construct validity, measurement properties and normative data in a large non-clinical sample. Br J Clin Psychol. 2004 Sep;43(Pt 3):245-65. doi: 10.1348/0144665031752934. PMID 15333231
- [Background] Azpiroz F, Guyonnet D, Donazzolo Y, Gendre D, Tanguy J, Guarner F. Digestive Symptoms in Healthy People and Subjects With Irritable Bowel Syndrome: Validation of Symptom Frequency Questionnaire. J Clin Gastroenterol. 2015 Aug;49(7):e64-70. doi: 10.1097/MCG.0000000000000178. PMID 25014236
- [Background] Guyonnet D, Schlumberger A, Mhamdi L, Jakob S, Chassany O. Fermented milk containing Bifidobacterium lactis DN-173 010 improves gastrointestinal well-being and digestive symptoms in women reporting minor digestive symptoms: a randomised, double-blind, parallel, controlled study. Br J Nutr. 2009 Dec;102(11):1654-62. doi: 10.1017/S0007114509990882. Epub 2009 Jul 22. PMID 19622191
- [Background] Marteau P, Guyonnet D, Lafaye de Micheaux P, Gelu S. A randomized, double-blind, controlled study and pooled analysis of two identical trials of fermented milk containing probiotic Bifidobacterium lactis CNCM I-2494 in healthy women reporting minor digestive symptoms. Neurogastroenterol Motil. 2013 Apr;25(4):331-e252. doi: 10.1111/nmo.12078. Epub 2013 Mar 11. PMID 23480238
- [Background] Rosas HD, Doros G, Bhasin S, Thomas B, Gevorkian S, Malarick K, Matson W, Hersch SM. A systems-level "misunderstanding": the plasma metabolome in Huntington's disease. Ann Clin Transl Neurol. 2015 Jul;2(7):756-68. doi: 10.1002/acn3.214. Epub 2015 May 28. PMID 26273688
- [Background] Boyle SH, Matson WR, Velazquez EJ, Samad Z, Williams RB Jr, Sharma S, Thomas B, Wilson JL, O'Connor C, Jiang W. Metabolomics analysis reveals insights into biochemical mechanisms of mental stress-induced left ventricular dysfunction. Metabolomics. 2015 Jun 1;11(3):571-582. doi: 10.1007/s11306-014-0718-y. PMID 25983674
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press; 1983.
- [Background] International Personality Item Pool: A Scientific Collaboratory for the Development of Advanced Measures of Personality Traits and Other Individual Differences [cited 2020]. Available from: http://ipip.ori.org/.
- [Background] Cohen S. Perceived stress in a probability sample of the United States. The social psychology of health. Thousand Oaks, CA, US: Sage Publications, Inc; 1988. p. 31-67.
- [Background] Addolorato G, Ancona C, Capristo E, Graziosetto R, Di Rienzo L, Maurizi M, Gasbarrini G. State and trait anxiety in women affected by allergic and vasomotor rhinitis. J Psychosom Res. 1999 Mar;46(3):283-9. doi: 10.1016/s0022-3999(98)00109-3. PMID 10193919
- [Background] Knight RG, Waal-Manning HJ, Spears GF. Some norms and reliability data for the State--Trait Anxiety Inventory and the Zung Self-Rating Depression scale. Br J Clin Psychol. 1983 Nov;22 (Pt 4):245-9. doi: 10.1111/j.2044-8260.1983.tb00610.x. PMID 6640176
- [Background] DHQ W-b. Diet History Questionnaire II & Canadian Diet History Questionnaire II: Web-based DHQ. 2021. Available from: https://epi.grants.cancer.gov/dhq2/.
- [Background] Goldberg LR. A broad-bandwidth, public domain, personality inventory measuring the lower-level facets of several five-factor models. In: Mervielde I, Deary I, De Fruyt F, Ostendorf F, editors. Personality Psychology in Europe. Tilburg, The Netherlands: Tilburg University Press; 1999. p. 7-28.
- [Background] Goldberg LR, Johnson JA, Eber HW, Hogan R, Ashton R, Cloninger CR, Gough HC. The International Personality Item Pool and the future of public-domain personality measures. Journal of Research in Personality. 2006; 40:84-96.
- [Background] IPIP. International Personality Item Pool: A Scientific Collaboratory for the Development of Advanced Measures of Personality Traits and Other Individual Differences. 2021. Available from: http://ipip.ori.org/.
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vag PR, Jacobs GA. Manual for the State-Trait Anxiety Inventory. 1983.

DOCUMENTS (1):
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT05026333/ICF_000.pdf